CLINICAL TRIAL: NCT00798863
Title: Video Assisted Submandibular Resection, Two Step Technique
Brief Title: Study Of The Safety And Efficacy Video Assisted Submandibular Gland Resection Using A New Two Step Technique
Acronym: VANSsubmand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Yasser Hamza, UAlexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VASS
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Submandibular Gland Resection
Keywords: submandibular gland; video assisted neck surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- operative group (Experimental): The patients of the group will have the operation of two step video assisted submandibular sialadenectomy.
  Interventions: Procedure: video assisted submandibular sialadenectomy

INTERVENTIONS:
Procedure: video assisted submandibular sialadenectomy — Step 1: A 15 to 20 mm skin incision is performed. The anterior part of the gland is then dissected off the mylohyoid muscle. The superficial part of the gland is dissected free. Now, the free superficial part of the gland is resected .Step 2: The scope is inserted into the wound to view the deeper part of the gland. The latter is dissected and removed after identifying the tendon of the digastric muscle, the hypoglossal nerve, the lingual nerve and the submandibular duct. The lingual nerve is released from its attachment to the gland. The submandibular duct is ligated using 3/0 vicryl. The deep part of the gland is extracted through the wound. Hemostasis is secured.
  Other Names: video assisted neck surgery

SUMMARY:
The study addresses a problem that face surgeons who perform key-hole surgery to resect the submandibular salivary gland. The problem is the narrow space available around that gland. This does not allow for a safe operation. The study aims to evaluate a new, two step resection technique, that should overcome this difficulty.

DETAILED DESCRIPTION:
The study included twelve adult patients suffering from chronic submandibular sialadenitis and indicated for sialadenectomy. The following exclusion criteria were adopted: Previous history of surgery or irradiation to the neck; History of abscess formation in the region; Patients having large, hard or fixed submandibular gland and where there was suspicion of malignancy. Laboratory work-up and ultrasound of the neck were obtained.All patients had video assisted submandibular sialadenectomy, using a "two step resection" technique as follows:Step 1: A 15 to 20 mm skin incision was performedThe edges of the wound are protected using a rubber cuff. The dissection is done using the harmonic scalpel in one hand and the suction spatula in the other hand. The anterior part of the gland is then dissected off the mylohyoid muscle. The plane of the dissected anterior pole of the gland is used as a guide. This plane is followed all around the gland until the whole superficial part of the gland is dissected free. Step 2: The retractors are adjusted to elevate the roof of the cavity created by removing the superficial part pf the gland. The scope is inserted into the wound to view the deeper part of the operative field. All nearby important structures are now identified and protected. The deep part of the gland is dissected and removed

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Has submandibular sialadenitis

Exclusion Criteria:

* Previous history of surgery or irradiation to the neck
* History of abscess formation in the region
* Patients having large, hard or fixed submandibular gland
* If there was suspicion of malignant submandibular tumour

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
incidence of complications after the operation | patients are examined for complications the next day of the operation

SECONDARY OUTCOMES:
operative time | operative time is calculated at the end of the operation
patient satisfaction with the cosmetic result of the operation | 12 weeks after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Hamza, A professor, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria University Hospitals, Alexandria, Alexandria Governorate, Egypt